CLINICAL TRIAL: NCT02380430
Title: Organisation PERiopératoire de l'anesthésie et de la Chirurgie Ambulatoire
Brief Title: Medical Management Survey : Organization of Perioperative Practices in Anesthesia and Ambulatory Surgery
Acronym: OPERA
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Société Française d'Anesthésie et de Réanimation (Other); Floralis (Industry)
Responsible Party: Sponsor
Other Study IDs: DCIC 1319
Record Dates: First submitted 2014-07-03; First posted 2015-03-05 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Surgery
Keywords: Ambulatory surgery; Pain management; Nausea and vomiting management; Questionnaire; Survey; Management
MeSH Terms: conditions — Agnosia; Nausea

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ambulatory surgery description: Medical questionnaire. Nausea and vomiting, pain, thromboprophylaxis description
  Interventions: Other: ambulatory surgery description

INTERVENTIONS:
Other: ambulatory surgery description — Medical questionnaire. Nausea and vomiting, pain, thromboprophylaxis description

SUMMARY:
In France, there are no precise data regarding perioperative organization of medical structure and care management of ambulatory surgical patients. Particularly, data on management of pain, nausea and vomiting, as well as venous thromboembolic, prevention and treatment are needed, in several groups of patients.

DETAILED DESCRIPTION:
This is a prospective epidemiological observationnal study involving a sample of 300 ambulatory surgical centers among 1000 french centers.

In a first step, a survey on the specific organization and care management of the structure will be carried out.

In a second step, data on the management of 3000 patients admitted in these structure will be performed. The will allow an analysis of practices in a selection of acts (which seem to be more frequent and more relevant). Data from three different questionnaires on pain management, PONV prevention and treatment and VTE prevention will be recorded for each patient.

ELIGIBILITY:
Inclusion Criteria:

* All patients managed for ambulatory surgery by medical structures during the two days of the survey.
* For the patient managed for specific ambulatory surgery by medical structures, a more detail survey will be conducted (if applicable). Specific surgery are :Oral surgery ( wisdom tooth extraction surgery), Knee arthroscopy, Abdominal wall surgery (including inguinal hernia surgery), Perianal surgery, Varicose veins surgery, Cholecystectomy/laparoscopy surgery, Lumpectomy, Uterine surgery, Hallux valgus, Hand surgery (except carpal tunnel surgery)

Exclusion Criteria: None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients managed for ambulatory surgery by medical structures.
Sampling Method: Non-Probability Sample
Enrollment: 2174 (Actual)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Description of amubalory surgery centers | Peri Operative Day 0
  Structure questionnaire
Description of organization and patient management | Peri Operative Day 0
  Management of ambulatory surgical patients using questionnaires including :
  Medical management questionnaire. Nausea and vomiting management questionnaire. Pain management questionnaire. Venous thromboprophylaxis management questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre ALBALADEJO, Professor, Principal Investigator — Pole anesthésie Réanimation - CHU de Grenoble; Jean Luc BOSSON, Professor, Study Director — Centre d'Investigation Clinique - Pavillon Taillefer - CHU de Grenoble
Locations (233):
- France (233):
  - Polyclinique de Deauville, Deauville, Cricquebœuf
  - Clinique Esquirol-Saint-Hilaire (CESH), Agen
  - Polyclinique du Parc Rambot, Aix-en-Provence
  - CHIC Alencon - Mamers, Alençon
  - CH Ales Cevennes, Alès
  - Centre Hospitalier - Altkirch, Altkirch
  - CH Ambert, Ambert
  - CHU - Amiens, Amiens
  - Groupe Santé Victor Pauchet, Amiens
  - Centre de la main - Angers, Angers
  - CHU Angers, Angers
  - Clinique Générale, Annecy
  - Hôpital Privé Antony, Antony
  - Centre Médico Chirurgical Wallerstein, Arès
  - CH Joseph Imbert, Arles
  - Polyclinique du Beaujolais, Arnas
  - CH - Aubagne, Aubagne
  - Hôpital Privé La Cassamance, Aubagne
  - CH - Auch, Auch
  - Centre hospitalier Henri Mondor d'Aurillac, Aurillac
  - CH Henri Duffaut, Avignon
  - Clinique St Antoine - Bastia, Bastia
  - CH - Bastia, Bastia
  - Centre Hospitalier de Bayeux, Bayeux
  - Clinique la Chataigneraie, Beaumont
  - Centre Hospitalier de Beaune, Beaune
  - CH Beaune, Beaune
  - CH - Béthune, Béthune
  - CH - Beziers, Béziers
  - Hopital Avicennes, Bobigny
  - Clinique du Cèdre, Bois-Guillaume
  - Clinique St Antoine, Bois-Guillaume
  - CHU - Groupe Hospitalier Pellegrin, Bordeaux
  - CHU Groupe Hospitalier Pellegrin 1, Bordeaux
  - Clinique Chirurgicale Bel Air 1, Bordeaux
  - Clinique chirurgicale Bel Air 2, Bordeaux
  - Clinique Convert, Bourg-en-Bresse
  - Clinique St Vincent de Paul, Bourgoin
  - Hôpital Instruction des Armées, Brest
  - CHRU Hôpital Morvan, Brest
  - CHU Brest, Brest
  - CHU - Caen, Caen
  - Fondation de la Misericorde - Caen, Caen
  - CHG - Cahors, Cahors
  - Clinique du Quercy, Cahors
  - Clinique Du Cambresis, Cambrai
  - Hôpital Privé Cannes Oxford, Cannes
  - Clinique du Parc, Castelnau-le-Lez
  - Polyclinique Sevigne, Cesson-Sévigné
  - CH Loire Vendée Océan, Challans
  - CH Chalon-sur-Saône, Chalon-sur-Saône
  - Pôle Santé Léonard de Vinci, Chambray-lès-Tours
  - Centre Hospitalier de Chartres, Chartres
  - CH - Chalons en Champagne, Châlons-en-Champagne
  - CH Châteauroux - Hôpital de Châteauroux, Châteauroux
  - CHP - Site de Cherbourg, Cherbourg
  - CH Clermont, Clermont-de-l'Oise
  - CHU Estaing, Clermont-Ferrand
  - APHP Cochin, Cochin
  - Groupe Hospitalier du Centre Alsace, Colmar
  - Polyclinique Saint Côme, Compiègne
  - Clinique des Cèdres, Cornebarrieu
  - Clinique de Flandre - Coudekerque Branche, Coudekerque-Branche
  - CH - Crest, Crest
  - CH - Denain, Denain
  - Hôpital Privé Saint-François, Désertines
  - Clinique Drevon, Dijon
  - CGFL Dijon, Dijon
  - CHU Dijon, Dijon
  - Clinique des Cèdres, Échirolles
  - CH Emile Durkheim - Epinal, Épinal
  - Clinique Saint-Dominique, Flers
  - CHI - Frejus Saint Raphaël, Fréjus
  - Polyclinique St Louis Languedoc Santé, Ganges
  - CHU - Hôpital Michallon, Grenoble
  - Groupe Hospitalier Mutualiste, Grenoble
  - Clinique de la Marche, Guéret
  - CH - Antibes Juan les pins, Juan-les-Pins
  - CH La Rochelle, La Rochelle
  - Centre hospitalier Ferdinand Grall, Landerneau
  - Clinique Sainte-Anne, Langon
  - Clinique de la Compassion, Langres
  - Centre Hospitalier Le Creusot-montceau, Le Creusot
  - Fondation Hôtel Dieu Le Creusot, Le Creusot
  - CH Hopital Jacques Monod, Le Havre
  - Clinique les ormeaux, Le Havre
  - Hopital privé de l'Estuaire, Le Havre
  - Centre de Chirurgie Abulatoire des Hauts d'Avignon, Les Angles
  - Clinique Lille Sud, Lesquin
  - CHRU Lille, Lille
  - Polyclinique du bois, Lille
  - Polyclinique La Louviere - Lille, Lille
  - Clinique Tous Vents, Lillebonne
  - CHU Dupuytren, Limoges
  - CH Lons, Lons
  - Centre Hospitalier de Bretagne Sud site Bodelio, Lorient
  - Clinique via domitia Pole de sante, Lunel
  - CH - Luneville, Lunéville
  - Clinique de la Sauvegarde, Lyon
  - HCL - Edouard Herriot, Lyon
  - HCL - Lyon Sud, Lyon
  - HCL Lyon - Croix-rousse, Lyon
  - Hôpital Privé Jean Mermoz, Lyon
  - Clinique Générale Marignane, Marignane
  - CHIC Marmande, Marmande
  - Clinique Baillis, Marmande
  - CH Lagny, Marne La Vallée
  - APHM - Hôpital de la Conception, Marseille
  - APHM Hôpital Sainte Marguerite, Marseille
  - Clinique de la Résidence du Parc, Marseille
  - Clinique Juge - Marseille, Marseille
  - Hôpital Européen - Marseille, Marseille
  - CH Mayotte, Mayotte
  - Polyclinique Val de Saone, Mâcon
  - CH-Meaux, Meaux
  - CH - Mende, Mende
  - Hopitaux Privés - Metz, Metz
  - Clinique de Meudon, Meudon-la-Forêt
  - CH Belfort Montbeliard, Montbéliard
  - CH du Forez - Montbrison, Montbrison
  - CH du Forez, Montbrison
  - Clinique Nouvelle du Forez, Montbrison
  - CH - Montelimar, Montélimar
  - CHU Arnaud de Villeneuve, Montpellier
  - CHU G. de Chauliac, Montpellier
  - CHU Lapeyronie, Montpellier
  - Clinique du Millenaire, Montpellier
  - ICM Institut Régional du cancer, Montpellier
  - Clinique de l'Esperance, Mougins
  - CH - Emile Muller, Mulhouse
  - Clinique Diaconnat Roosevelt, Mulhouse
  - Clinique Diaconnat-Fonderie, Mulhouse
  - Centre Chirurgical Emile Gallé - SINCAL, Nancy
  - CHU - Nancy, Nancy
  - Polyclinique de Gentilly, Nancy
  - CHU Nantes, Nantes
  - Clinique Hartmann, Neuilly-sur-Seine
  - Clinique Pierre Cherest, Neuilly-sur-Seine
  - Clinique Sainte Isabelle, Neuilly-sur-Seine
  - CHAN - Nevers, Nevers
  - CH Georges Renon - Niort, Niort
  - Polyclinique Inkermann, Niort
  - CHU Caremeau, Nîmes
  - Polyclinique Grand Sud, Nîmes
  - Centre Hospitalier de Nogent le Rotrou, Nogent-le-Rotrou
  - CHIC - Noyon, Noyon
  - CHIC Noyon, Noyon
  - Polyclinique Mutualiste Malartic, Ollioules
  - CHR Orléans, Orléans
  - Clinique Sainte Marie, Osny
  - CH Paray, Paray
  - APHP - Ambroise Pare, Paris
  - APHP - Necker, Paris
  - APHP Hôpital Trousseau, Paris
  - APHP Kremlin Bicetre, Paris
  - APHP Lariboisière, Paris
  - Aphp-Hegp, Paris
  - APHP-St Antoine, Paris
  - APHP-Tenon, Paris
  - CH National d'Ophtalmologie - les quinze vingts, Paris
  - Clinique Ambroise Pare, Paris
  - Clinique Arago, Paris
  - Clinique st Jean de Dieu, Paris
  - Fondation Ophtalmologique Rothschild, Paris
  - Institut Mutualiste Montsouris, Paris
  - Polyclinique de Navarre, Pau
  - Clinique Mutualiste Catalane, Perpignan
  - Clinique Mutualiste de Pessac, Pessac
  - Hôpital Privé Saint-Martin, Pessac
  - Clinique du Ter, Ploemeur
  - CH Poissy, Poissy
  - Clinique St Louis, Poissy
  - CHU - Poitiers, Poitiers
  - Clinique de l'Atlantique, Puilboreau
  - CHIC Cornouaille, Quimper
  - CH Rambouillet, Rambouillet
  - CH - arrondissement de Montreuil, Rang-du-Fliers
  - Centre Hospitalier de Redon, Redon
  - Hôpital Robert Debré- CHU de Reims, Reims
  - CH - Remiremont, Remiremont
  - CHU - Hôpital Sud - Rennes, Rennes
  - CHU - Pontchaillou - Rennes, Rennes
  - Centre Hospitalier Guy Thomas de Riom, Riom
  - Clinique du Renaison, Roanne
  - CH - Rodez, Rodez
  - CHU Rouen, Rouen
  - CRLCC Henri Becquerel, Rouen
  - Clinique Pasteur - Royan, Royan
  - Clinique de l'Alliance, Saint-Cyr-sur-Loire
  - CHU Félix Guyon, Saint-Denis
  - CHU Hôpital Nord, Saint-Etienne
  - CHU St Etienne - Hôpital Nord, Saint-Etienne
  - Clinique Mutualiste Chirurgicale, Saint-Etienne
  - CH Comminges Pyrenees, Saint-Gaudens
  - CH Saint-Germain-en-Laye, Saint-Germain-en-Laye
  - CH - St-Jean d'Angely, Saint-Jean-d'Angély
  - Clinique Gaston Metivet, Saint-Maur
  - CH - St Omer, Saint-Omer
  - Clinique Des landes, Saint-Pierre-du-Mont
  - CH - St Quentin, Saint-Quentin
  - Clinique Vignoli, Salon-de-Provence
  - CH Seclin, Seclin
  - CH-Seclin, Seclin
  - Centre Hospitalier de Semur-en-Auxois, Semur-en-Auxois
  - CHIC Bassin de Thau - Sete, Sète
  - Clinique Saint Christophe Courlancy, Soissons
  - Institut Ophtalmique, Somain
  - Clinique Diaconesses, Strasbourg
  - Clinique Sainte Odile, Strasbourg
  - CHU de Strasbourg, Strasbourg
  - Clinique Orangerie, Strasbourg
  - CH Saint-Jacques, Thann
  - CH - Toul, Toul
  - CH Toulon, Toulon
  - CHU - Toulouse, Toulouse
  - Hopital Joseph Ducuing, Toulouse
  - Institut Claudius Regaud, Toulouse
  - Polyclinique du Parc, Toulouse
  - CHRU Tours, Tours
  - Centre Hospitalier de Troyes, Troyes
  - CH - Valence, Valence
  - Hôpital privé Océane, Vannes
  - Centre Hospitalier Bretagne Atlantique site de Vannes, Vannes
  - CH - Verdun, Verdun
  - Polyclinique la pergola, Vichy
  - Centre Hospitalier du Vierzon, Vierzon
  - CH - Villefranche sur Saone, Villefranche-sur-Saône
  - Clinique de Villeneuve d'Ascq, Villeneuve-d'Ascq
  - Centre Hospitalier Saint-Cyr- Villeneuve sur Lot, Villeneuve-sur-Lot
  - CH Villeneuve sur Lot, Villeneuve-sur-Lot
  - Clinique Notre Dame, Vire
  - CH - Voiron, Voiron
  - Hôpital Privé du Val d'Yerres, Yerres

REFERENCES:
- [Background] Clergue F, Auroy Y, Pequignot F, Jougla E, Lienhart A, Laxenaire MC. [Anesthesia in France in 1996. Results of a study of the French Society of Anesthesia and Resuscitation]. Chirurgie. 1999 Apr;124(2):115-21. doi: 10.1016/s0001-4001(99)80053-1. No abstract available. French. PMID 10349747
- [Background] Clergue F, Auroy Y, Pequignot F, Jougla E, Lienhart A, Laxenaire MC. French survey of anesthesia in 1996. Anesthesiology. 1999 Nov;91(5):1509-20. doi: 10.1097/00000542-199911000-00045. PMID 10551604
- [Background] Lienhart A, Auroy Y, Clergue F, Laxenaire MC, Pequignot F, Jougla E. [Anesthetics and transfusion practices]. Ann Fr Anesth Reanim. 1998;17(11):1374-86. doi: 10.1016/s0750-7658(99)80050-1. No abstract available. French. PMID 9972365
- [Derived] Aubrun F, Ecoffey C, Benhamou D, Jouffroy L, Diemunsch P, Skaare K, Bosson JL, Albaladejo P. Perioperative pain and post-operative nausea and vomiting (PONV) management after day-case surgery: The SFAR-OPERA national study. Anaesth Crit Care Pain Med. 2019 Jun;38(3):223-229. doi: 10.1016/j.accpm.2018.08.004. Epub 2018 Oct 16. PMID 30339892